CLINICAL TRIAL: NCT00333242
Title: Hyperalgesia in Methadone Patients: Can it be Treated?
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Margaret (Peggy) Compton RN PhD, UCLA School of Nursing
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01DA015463-04 (NIH)
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2008-08

CONDITIONS: Opioid-induced Hyperalgesia
Keywords: Pain; opioid; hyperalgesia; methadone
MeSH Terms: conditions — Pain; Hyperalgesia | interventions — Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Drug: dextromethorphan — dextromethorphan PO titrated to 480 mg/day x 5 weeks

SUMMARY:
In the proposed study, we will build upon our previous studies validating and characterizing hyperalgesia in MM samples to explore it's underlying mechanism from a pharmacological perspective. Utilizing a double-blind, placebo-controlled designs, the proposed work will evaluate the ability of dextromethorphan , an N-methyl-D-aspartate (NMDA)-antagonists to diminish or reverse the opioid-induced hyperalgesia complicating the pain states suffered by MM patients. Specifically, in a sample of MM patients, dextromethorphan, theorized to interfere with the development of opioid-induced hyperalgesia will be evaluated for its ability to ameliorate or diminish the opioid-induced hyperalgesia in these patients as reflected by changes on pain threshold and tolerance to both cold-pressor and electrical pain, at peak and trough methadone blood levels. The results of this work will not only provide pharmacologic insight into the mechanisms underlying poor pain tolerance in this at-risk population, but also direction for the medical management of pain complicated by opioid-induced hyperalgesia.

DETAILED DESCRIPTION:
Addressing the undertreatment of clinical pain has become a national priority, with a central goal being to identify effective interventions for those subgroups of patients most at risk for suffering unrelieved pain (NIH Program Announcement PA-01-115). In fact, the undertreatment of pain was recently ruled a form of patient abuse with a California court awarding one million dollars in damages to the family of such a patient. Novel data accumulated by our investigative group has shown that patients maintained on the mu-opioid agonist, methadone, for the treatment of addiction, are significantly hyperalgesic to cold-pressor experimental pain as compared to normal controls. This diminished pain tolerance, in addition to the contextual prohibitions associated with providing known opioid addicts with opioid analgesics, makes them a population uniquely vulnerable to the undertreatment of pain. Unfortunately, little is known about how to best manage the pain suffered by the over 120,000 methadone-maintained (MM) patients in this country, in part because the hyperalgesia they suffer appears to be akin to neuropathic pain and opioid-induced.

In the proposed series of studies, the Principal Investigator (a first-time R01 applicant) will build upon her previous studies validating and characterizing hyperalgesia in MM samples to explore it's underlying mechanism from a pharmacological perspective. Utilizing slightly different double-blind, placebo-controlled designs, the proposed work will evaluate the ability of three classes of medication (N-methyl-D-aspartate (NMDA)-antagonists, adjuvant anticonvulsant analgesics, and novel opioid analgesics) to diminish or reverse the opioid-induced hyperalgesia complicating the pain states suffered by MM patients. Specifically, in a sample of MM patients, (1) dextromethorphan, which interferes with the development of opioid-induced hyperalgesia, (2) gabapentin, which has proven efficacy in treating neuropathic pain, and (3) oxycodone, which has novel opioid activity, will each be evaluated for its ability to ameliorate or diminish the opioid-induced hyperalgesia in these patients as reflected by changes on pain threshold and tolerance to both cold-pressor and electrical pain, at peak and trough methadone blood levels. The results of this work will not only provide pharmacologic insight into the mechanisms underlying poor pain tolerance in this at-risk population, but also direction for the medical management of pain complicated by opioid-induced hyperalgesia.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: Potential participants must:

  1. Be between the ages of 18 and 55 years of age.
  2. Fulfill DSM-IV criteria for opiate dependence.
  3. Be compliant in MM treatment and on a stable dose of methadone x 6 weeks.
  4. Be in good physical health or in the case of a medical condition needing ongoing treatment, be in the care of a physician who is willing to take responsibility for such treatment. The same conditions apply in cases of patients with a psychiatric disorder needing ongoing treatment.
  5. Be agreeable to and capable of signing an informed consent.

Exclusion Criteria:

* Exclusion Criteria: Potential participants must not:

  1. Have known sensitivity to dextromethorphan, gabapentin or oxycodone.
  2. Be dependent on alcohol, benzodiazepine or other drugs of abuse (except nicotine).
  3. Have any acute medical condition that would make participation medically hazardous, (e.g., acute hepatitis, unstable cardiovascular disease, liver or renal disease) or have liver enzyme values (AST or ALT) greater than 5 times normal range.
  4. Be acutely psychotic, severely depressed and in need of inpatient treatment, or an immediate suicide risk.
  5. Have a neurological or psychiatric illness (i.e., peripheral neuropathy, schizophrenia, neuropathic pain, Raynaud's disease, urticaria,) that would affect pain responses.
  6. Be currently taking analgesic medication (opioid or otherwise) for a painful condition on a regular basis.
  7. Be a nursing or pregnant female. Female of childbearing potential must agree to use a medically acceptable method of birth control, (e.g. oral contraceptives, barrier (diaphragm or condom) with or without spermicide, levonorgestrel implant, intra-uterine progesterone contraceptives system, medroxyprogesterone acetate contraceptive injection) or to complete abstinence. Females who become pregnant during the course of the study will be dropped from the study.
  8. Have a current or past history of high blood pressure, heart disease, stroke or currently have a pacemaker.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2002-09; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Pain tolerance | 6 week

SECONDARY OUTCOMES:
Pain threshold | 6 week

CONTACTS AND LOCATIONS:
Overall Officials: Margaret A Compton, RN, PhD, Principal Investigator — UCLA School of Nursing
Locations (1):
- UCLA School of Nursing, Los Angeles, California, United States